CLINICAL TRIAL: NCT05082675
Title: A Phase-II Study Comparing Non-Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation Following Autologous Transplantation to Autologous Transplantation Alone in Multiple Myeloma
Brief Title: Stem Cell Translpantation in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Society for Blood and Marrow Transplantation (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMAM2000
Record Dates: First submitted 2021-09-21; First posted 2021-10-19 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2021-10

CONDITIONS: Multiple Myeloma
Keywords: myeloma; HLA-matched; autologous; allogeneic; transplant
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: Patients with an HLA-identical sibling donor were allocated to the auto-allo arm (n = 108) and patients without a matched sibling donor were allocated to the auto arm (n = 249)

ARMS (2):
- auto/RICallo treatment arm (Experimental): Patients with an HLA-identical sibling donor were allocated to the auto-allo arm (n = 108)
  Interventions: Procedure: HLA Matched allogeneic transplant
- auto arm (Active Comparator): patients without a matched sibling donor were allocated to the auto arm (n = 249). Single (n = 145) or tandem (n = 104)
  Interventions: Procedure: HLA Matched allogeneic transplant

INTERVENTIONS:
Procedure: HLA Matched allogeneic transplant

SUMMARY:
The purpose of this study is to determine whether autologous transplantation (using the patient's own stem cells from the blood), followed by non-myeloablative (i.e. less intense) allogeneic transplantation (where the blood stem cells from a sibling donor are used for the transplantation) improves the outcome in patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
This trial includes a natural (no available HLA-identical sibling donor) control arm. Patients with newly diagnosed multiple myeloma without a sibling are initially treated with conventional chemotherapy followed by conventional single or double autologous transplant (PBSCT). Data from this group is used as part of the control group.

Eligible patients with one or more sibling are offered to participate in the main trial arm. Those who decline are asked to consider taking part in the control group (autograft only).

Patients consenting to participate in the main study first receive the PBSCT, followed by the HLA-matched non-myeloablative allograft (matched for HLA -A, -B, -C, -DRB1).

All study patients receive four to six cycles of VAD (or alternative regimens specified in protocol) before PBSCT as first line treatment. Study entry starts at the time of starting conditioning for autologous transplantation. The search for an identical sibling donor begins as soon as the patient has consented to participate in the study.

The allograft is performed when the patient has restored their marrow function but no earlier than 3 months following PBSCT.

The aim is to demonstrate a difference in outcome (progression free survival, transplant related mortality, relapse rate, and survival).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Stage-II and III multiple myeloma (According to Durie and Salmon classification)
* Age under 70 years
* Life expectancy over 3 months
* Patients must be able to give informed consent

Exclusion Criteria:

* Serious concomitant medical disease which would limit life span or the ability to tolerate chemotherapy
* Severe cardiac failure (ejection fraction <40%)
* Impairment of renal function at diagnosis is not per se reason for exclusion but patients with severe impaired renal function (GFR <50 ml/min) after initial VAD (or VAD like) induction treatment are excluded
* Severe impairment of liver function (bilirubin >2 times upper limit of normal)
* Pregnant or lactating women
* Other major organ system dysfunction (GI, neurological, psychiatric dysfunction) that impairs tolerance of therapy or prolong hematological recovery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2001-09; Primary Completion 2011-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  Progression free survival

SECONDARY OUTCOMES:
Transplant related mortality | 5 years
  Transplant related mortality
Complete hematological and molecular remission rate | 5 years
  Complete hematological and molecular remission rate
Relapse rate | 5 years
  Relapse rate
Survival | 5 years
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Bo Björkstrand, MD, Study Chair — Huddinge University Hospital
Locations (24):
- Medizinische Universität Wien, Vienna, Austria
- Québec, Canada
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Herlev Hospital, Herlev
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
  - Turku University, Turku
- CHU Lapeyronie, Montpellier, France
- Germany (2):
  - University of Heidelberg, Heidelberg
  - University of Leipzig, Leipzig
- Italy (5):
  - Ospedale Ferrarotto, Catania
  - Ospedale di Careggi, Florence
  - University of Milano, Milan
  - Uni. Modena, Policlinico, Modena
  - IRCCS, Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Norway (3):
  - Rikshospitalet, Oslo
  - Tromsø
  - Trondheim
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Huddinge University Hospital, Huddinge
  - Stockholm
  - University Hospital, Uppsala
- University Faculty of Medicine, Ankara, Turkey (Türkiye)
- Royal Marsden Hospital, London, United Kingdom

REFERENCES:
- See also: Sponsor's website — http://www.ebmt.org